CLINICAL TRIAL: NCT01143974
Title: Trial of Pemetrexed in Combined With Cisplatin for the Treatment of Advanced Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Associate chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-008
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Locally Advanced Malignant Neoplasm
Keywords: progress free survival; response rate; safety
MeSH Terms: interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PC Regimen (Experimental)
  Interventions: Drug: pemetrexed plus cisplatin

INTERVENTIONS:
Drug: pemetrexed plus cisplatin — pemetrexed 500mg/m2 plus cisplatin 80mg/m2 on day1 of each 21 day cycle, until progression
  Other Names: Alimta

SUMMARY:
For patients resistant to enthrycycline and taxanes, there is no standard regimen. Pemetrexed alone had certain efficacy in treatment of advance breast cancer. Platin was also a effective drug for advanced breast cancer. The combination of these two drug may have a synergy with each other in treatment of advanced breast cancer.

DETAILED DESCRIPTION:
combination of pemetrexed and cisplatin to treat advanced breast cancer. Previous regimen no more than 3 which including enthrycycline and taxanes(paclitaxel and/or docetaxel)

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Resistant to enthracycle and taxanes
* Has measurable disease

Exclusion Criteria:

* Has more than 3 previous chemotherapy regimens

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
PFS (progression free survival) | 2 Years

SECONDARY OUTCOMES:
Safety | 2 years
  Assessing for Hematology and Non-hematology toxicities, including all SAEs.
Response Rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, M.D., Study Chair — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute & Hospital. Chinese Academy of Medical Sciences, Beijing, China